CLINICAL TRIAL: NCT02951000
Title: Platysma Trial - a Randomized Controlled Trial of Platysma Suturing Versus no Sutures for Wound Closure After Primary Thyroid Surgery
Brief Title: Platysma Trial - Platysma Suturing Versus no Sutures for Wound Closure After Primary Thyroid Surgery
Acronym: Platysma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLA1
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-10

CONDITIONS: Thyroid Disease
Keywords: thyroidectomy; postoperative pain; wound healing
MeSH Terms: conditions — Thyroid Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- platysma suture (Active Comparator): running suture of the platysma with 3/0 polyglactin
  Interventions: Procedure: platysma suture
- no platysma suture (Active Comparator): no platysma suture
  Interventions: Procedure: no platysma suture

INTERVENTIONS:
Procedure: platysma suture
  Arms: platysma suture
Procedure: no platysma suture
  Arms: no platysma suture

SUMMARY:
Influence of the platysma suture on postoperative pain and wound healing.

DETAILED DESCRIPTION:
Does a running platysma suture after primary thyroid resection alter direct postoperative pain, wound healing and long term cosmetic results.

Primary outcome measure is if the lack of a platysma-Suture decreases the postoperative pain (detected by the visual pain score 0-10) and reduces the pain medication (detected by the cumulative NSAID and opioid treatment per patient). The second Question to be answered is if the cosmetic scar result (detected by the Patient and Observer Scar Assessment Score) 6 month after thyroidectomy is better in the intervention group (no Platysma-Suture) or not.

ELIGIBILITY:
Inclusion Criteria:

* primary thyroid surgery

Exclusion Criteria:

* previous neck surgery
* application of wound drainages
* preoperative diagnosed malignancy
* surgical extension beyond thyroid resection (e.g. lymphadenectomy)
* preexisting coagulopathy
* preexisting chronic pain syndromes
* preexisting dependency on pain reliefs
* preexisting disorders in wound healing (e.g. diabetes mellitus)
* intolerance to any study medication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Pain at morning of the first postoperative day
  visual analogue pain scale (0-10)

SECONDARY OUTCOMES:
wound infection | within 14 days postoperative
  wound infections needing antibiotics or reintervention
scar cosmesis | 6 months after surgery
  scar cosmesis according to patient and observer scar assessment scale (POSAS)
Postoperative Pain | Pain 6h after surgery, at the morning of the second postoperative day, 14 days after surgery
  visual analogue pain scale (0-10)
Cervical Seroma/Hematoma | 14 days after surgery
  clinical apparent swelling verified by ultrasound
Disorders of the functional anatomy of the neck | At six months postoperative
  New onset of clinically described swallowing problems and reduced depression of the corners of the mouth

CONTACTS AND LOCATIONS:
Overall Officials: Sven Müller, MD, Principal Investigator — University Tuebigen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Senne M, Zein R, Falch C, Kirschniak A, Koenigsrainer A, Muller S. Randomized clinical trial of platysma muscle suture versus no suture for wound closure after thyroid surgery. Br J Surg. 2018 May;105(6):645-649. doi: 10.1002/bjs.10829. Epub 2018 Mar 26. PMID 29579320